CLINICAL TRIAL: NCT01773681
Title: Novel Imaging Markers for Rheumatoid Arthritis
Acronym: NIMRA
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: UCBCelltech
Record Dates: First submitted 2013-01-16; First posted 2013-01-23 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood sample will be collected and stored at Mary Nakamura's lab at the SF VAMC for future studies.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Cimzia — For the loading phase, it consists of the first 3 doses. During the loading phase, the recommended dose of Cimzia for adults with rheumatoid arthritis is 400mg initially followed by 400mg again at week 2 and week 4. A 400mg dose requires 2 subcutaneous injection of 200mg; the injections should occur at separate sites in the thigh or abdomen.
  After the loading dose, will be follow with 200mg every other week. The injection should occur at either the thigh or abdomen.
Device: Magnetic Resonance Imaging (MRI) — MRI of the dominant wrist, before, during and after the gadolinium contrast injection will be acquired. The dose of the gadolinium agent for this study is 0.1mmol/kg body weight. This gadolinium contrast agent will increase the image contrast in the joints in the wrist and surrounding tissues and will make the MRI pictures stand out better.
Device: High-resolution peripheral quantitative computed tomography (HR-pQCT) — HR-pQCT scan of the hand and wrist will be acquired to look at the bone quality. The scan uses special x-ray equipment to make detailed pictures of bone structure.
  Other Names: Scanco

SUMMARY:
The purpose of this study is to use magnetic resonance imaging (MRI) and high-resolution peripheral quantitative computed tomography (HR-pQCT) techniques to look at the damage and disease activity progression in the hand and wrist joints of patients with rheumatoid arthritis.

The central hypothesis is that ongoing erosions and cartilage loss in rheumatoid arthritis are due to persistent inflammation, which is poorly detected by clinical examination and markers of systemic inflammation.

ELIGIBILITY:
The inclusion criteria for all patients to be enrolled are:

* RA by 2010 ACR classification criteria
* Age ≥ 18 years at enrollment
* Ability to give consent and follow the study protocol
* Prednisone permitted in doses ≤10 mg daily
* Women of reproductive potential must agree to use an acceptable method of birth control during treatment

Additional inclusion criteria for group I:

* DAS28 ≤ 3.2 during the last 2-months prior to the baseline visit
* On MTX at a stable dose for > 8 weeks prior to the baseline visit
* No biologic therapy during the past 6-months prior to the baseline visit
* No anticipated biologic therapy

Additional inclusion criteria for group II:

* DAS28 > 3.2
* No biologic therapy during the past 6-months prior to the baseline visit
* Scheduled to initiate anti-TNF therapy using CIMZIA

Exclusion Criteria for all patients to be enrolled are:

* Any psychiatric disorder that prevents the subject from providing informed consent
* Inability or unwillingness to follow the protocol
* Estimated glomerular filtration rate (eGFR, calculated based on serum creatinine) < 60 ml/min/1.72m2
* Known allergy or hypersensitivity to any study products (including gadolinium)
* History of injury or surgery of the wrist and hand to be scanned
* Inability to place non-dominant hand appropriately for imaging
* History of claustrophobia; inability to tolerate MRI and other contraindication of MRI
* Pregnancy or breast-feeding
* Diabetes mellitus requiring insulin therapy
* Prednisone dose > 10 mg/day (or equivalent dose of another corticosteroid) within 1 month of baseline visit
* Any investigational agent within the earlier of 4 weeks or 5 half-lives prior to randomization
* Any biologic therapy within 6-month prior to the baseline visit
* Any condition or treatment, which in the opinion of the investigator, places the subject at an unacceptable risk as a participant in the study

Additional exclusion criteria for Group II:

* Chronic or persistent infection including but not limited to human immunodeficiency virus [HIV], hepatitis B, hepatitis C, listeriosis, TB, or other opportunistic infection)
* Active infection or severe infections requiring hospitalization or treatment with intravenous (IV) antibiotics, IV antivirals, or IV antifungals within 30 days prior to baseline visit, or oral antibiotics, oral antivirals, or oral antifungals within 14 days prior to baseline visit
* Receipt of a live vaccine within 4 weeks prior to baseline visit
* History of malignancy within the past 5 years other than treated localized carcinoma in situ of the cervix or adequately treated non-metastatic squamous or basal cell skin carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the UCSF RA Cohort by Drs. John Imboden and Jonathan Graf at SFGH and UCSF Medical Center RA Clinics.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
To better understand how Cimzia and methotrexate affect the damage and disease activity progression in the hand and wrist of patients with rheumatoid arthritis | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojuan Li, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF - China Basin Imaging Center, San Francisco, California, United States